CLINICAL TRIAL: NCT03430232
Title: A First-in-Human, Randomized, Double-blind, Placebo-controlled Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of STR-324 in Healthy Subjects
Brief Title: First-In-Human PainCart Study for STR-324
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stragen France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STR-324-CL-039; 2014-002402-21 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-02-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: For part I: crossover model For part II: parallel model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part I (Panel 1): STR-324 or placebo (Experimental): Subjects will receive STR-324 dose level 1, 3, 5, 7 or placebo as a short infusion according to randomization.
  Interventions: Drug: Placebo; Drug: STR-324 Dose Level 1; Drug: STR-324 Dose Level 3; Drug: STR-324 Dose Level 5; Drug: STR-324 Dose Level 7
- Part I (Panel 2): STR-324 or placebo (Experimental): Subjects will receive STR-324 dose level 2, 4, 6, 8 or placebo as a short infusion according to randomization.
  Interventions: Drug: Placebo; Drug: STR-324 Dose Level 2; Drug: STR-324 Dose Level 4; Drug: STR-324 Dose Level 6; Drug: STR-324 Dose Level 8
- Part II (Panel 1): STR-324 or placebo (Experimental): Subjects will receive STR-324 dose level A or placebo as a long infusion according to randomization.
  Interventions: Drug: STR-324 Dose Level A; Drug: Placebo
- Part II (Panel 2): STR-324 or placebo (Experimental): Subjects will receive STR-324 dose level B or placebo as a long infusion according to randomization.
  Interventions: Drug: STR-324 Dose Level B; Drug: Placebo
- Part II (Panel 3): STR-324 or placebo (Experimental): Subjects will receive STR-324 dose level C or placebo as a long infusion according to randomization.
  Interventions: Drug: STR-324 Dose Level C; Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Short infusion of the solution for intravenous administration, Sodium Chloride 0.9%
  Arms: Part I (Panel 1): STR-324 or placebo; Part I (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level 1 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 1): STR-324 or placebo
Drug: STR-324 Dose Level 2 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level 3 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 1): STR-324 or placebo
Drug: STR-324 Dose Level 4 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level 5 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 1): STR-324 or placebo
Drug: STR-324 Dose Level 6 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level 7 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 1): STR-324 or placebo
Drug: STR-324 Dose Level 8 — Short infusion of a solution for intravenous administration
  Arms: Part I (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level A — Long infusion of a solution for intravenous administration
  Arms: Part II (Panel 1): STR-324 or placebo
Drug: STR-324 Dose Level B — Long infusion of a solution for intravenous administration
  Arms: Part II (Panel 2): STR-324 or placebo
Drug: STR-324 Dose Level C — Long infusion of a solution for intravenous administration
  Arms: Part II (Panel 3): STR-324 or placebo
Drug: Placebo — Long infusion of the solution for intravenous administration, Sodium Chloride 0.9%
  Arms: Part II (Panel 1): STR-324 or placebo; Part II (Panel 2): STR-324 or placebo; Part II (Panel 3): STR-324 or placebo

SUMMARY:
This is an interventional, first-in-man study, double-blind, placebo-controlled, two-part, ascending doses study to investigate the safety, tolerability and efficacy of STR-324 infusions in healthy volunteers.

DETAILED DESCRIPTION:
Part I : ascending doses of short lasting infusion Part II : ascending doses of long lasting infusion

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure
* Healthy male subjects, 18 to 45 years of age, inclusive at screening.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive at screening, and with a minimum weight of 50 kg.
* All males must practice effective contraception during the study and be willing and able to continue contraception for at least 90 days after their last dose of study treatment.
* Has the ability to communicate well with the Investigator in the Dutch language and willing to comply with the study restrictions.

Exclusion Criteria:

* Evidence of any active or chronic disease or condition that could interfere with, or for which the treatment of might interfere with, the conduct of the study, or that would pose an unacceptable risk to the subject in the opinion of the investigator
* Subject with clinically significant abnormalities in blood pressure, heart rate, ECG recording and laboratory parameters
* Abnormal renal function (eGFR (MDRD) < 60 mL/min/1.73m2).
* Previous history of seizures or epilepsy.
* Acute disease state (e.g. nausea, vomiting, fever, or diarrhea) within 7 days before the first study day.
* Positive Hepatitis B surface antigen (HBsAg), Hepatitis B antibodies, Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab)
* Use of any medications (prescription or over-the-counter [OTC]), within 14 days of study drug administration, or less than 5 half-lives (whichever is longer).
* Use of any vitamin, mineral, herbal, and dietary supplements within 7 days of study drug administration, or less than 5 half-lives (whichever is longer).
* Participation in an investigational drug or device study within 3 months prior to first dosing.
* History of abuse of addictive substances or current use of substances (alcohol, illegal substances)
* Positive test for drugs of abuse or alcohol breath test at screening or pre-dose.
* Any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Loss or donation of blood over 500 mL within three months prior to screening
* Any current, clinically significant, known medical condition in particular any existing conditions that would affect sensitivity to cold or pain

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: number of subjects who experience (serious) treatment emergent adverse events, potential clinically changes in vital signs, ECG, holter, physical examinations, laboratory tests and urine production | Day 7 (+/- 2 days) post dosing

SECONDARY OUTCOMES:
Parts I and II: Maximum plasma concentration (Cmax) | Up to 24 hours for Part I and up to 52 hours for Part II
Parts I and II:Time to maximum plasma concentration (Tmax) | Up to 24 hours for Part I and up to 52 hours for Part II
Parts I and II: Area under the plasma concentration-time curve from zero to infinity(AUC0-inf) | Up to 24 hours for Part I and up to 52 hours for Part II
Parts I and II: Area under the plasma concentration-time curve from zero to the last measured concentration above the limit of quantification (AUC0-last) | Up to 24 hours for Part I and up to 52 hours for Part II
Parts I and II: Terminal disposition rate constant (λz) with the respective half-life (t½) | Up to 24 hours for Part I and up to 52 hours for Part II
Parts I and II: Amount excreted in urine in 24 hours | Up to 24 hours for Part I and up to 72 hours for Part II
Parts I and II: Thermal Pain | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Electrical pain Stair and Burst | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Pressure Pain | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Cold Pressor | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Conditioned Pain Modulation Response (change from electrical stair pre- and post-cold pressor) | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Visual Analogue Scale Bond & Lader | Up to 5 hours for part I and up to 56 hours for part II
Parts I and II: Visual Analogue Scale Bowdle | Up to 5 hours for part I and up to 56 hours for part II
Part II only: Saccadic eye movement | Up to 56 hours
Part II only: Smooth pursuit eye movement | Up to 56 hours
Part II only: Adaptive tracking | Up to 56 hours
Part II only: Body sway | Up to 56 hours
Part II only: N-Back | Up to 56 hours
Part II only: Pharmaco-EEG: power | Up to 56 hours
Part II only: Pupillometry | Up to 56 hours
Part II only: 49-item Addiction Center Research Inventory | Up to 60 hours
Part II only: Bowel Function Index | Up to day 7
Part II - Groups 2 and 3 only: Thermal pain (Normal skin and erythema skin - UVB) | Up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHDR, Leiden, Netherlands